CLINICAL TRIAL: NCT01653691
Title: Tunable-Dye Laser Therapy to Ameliorate Hypertrophic Scarring in Burned Children
Brief Title: Laser Therapy for Treating Hypertrophic Burn Scars in Children
Acronym: LaserTherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Mattias Donelan, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-P-002148
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Burn Scars
Keywords: Pediatric; Burns; Scars; Pulse Dye laser
MeSH Terms: conditions — Burns; Cicatrix | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulse Dye Laser, burn scars (Active Comparator): A scar will be located on the study subject's torso or thigh and divided in half. Some subjects will receive laser to both sides of their scar, while others will not receive any intervention to one side and laser to the other side. Each side will be evaluated during outpatient visits. 12 months after treatment is completed, 2 burn experts will rate each side of the scar without knowing its treatment.
  Interventions: Procedure: Pulse-Dye Laser
- No treatment to half of scar (Sham Comparator): A scar on the child's torso or thigh will be divided in half. One side will receive laser treatment and the other half will receive laser or sham treatment.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Pulse-Dye Laser — Laser therapy will be applied to either one half or both halves of the subject's burn scar. Laser will be re-applied every 4-6 weeks for a total of 3 administrations.
  Other Names: Candela V-Beam tunable dye laser.
  Arms: Pulse Dye Laser, burn scars
Procedure: Sham — No treatment to one side of subject's scar.
  Other Names: No treatment
  Arms: No treatment to half of scar

SUMMARY:
Pulse-dye laser therapy has been used to treat the redness, tightness and discomfort of hypertrophic scars resulting from burn injuries. To date the effectiveness of laser therapy on children's burned scars has not been measured.

DETAILED DESCRIPTION:
In this study we hope to answer an important question in pediatric burn care: what are the techniques whereby tunable-dye laser neo-vessel ablation is optimally employed to ameliorate hypertrophic scars resulting from burn injuries in children? Hypertrophic scarring is considered an adverse wound healing event that results in abnormal scar formation. This scarring process is associated with pruritis and discomfort and can interfere with function and aesthetics. Topical creams, massage, stretching and pressure are used as standard treatments of burn scar formation. With the child serving as their own control, we want to objectively measure the impact of PDL on burn scars in children. Variables of timing of application, duration and number of sessions will all be collected.

ELIGIBILITY:
Inclusion Criteria:

* subjects 9 years and older to 21 years of age or younger with a second degree burn with erythema and the potential for hypertrophic scarring to the thigh and or trunk.
* subject is clinically stable within 3 months of the burn injury.
* burn size of at least 15cm2 and able to be divided into equivalent halves (divided along line of tension). Equivalent orientation distance from mobil joint with regard to history,physical findings, proximity to tension producing forces and orientation.
* subjects in acute phase of burn injury generally less than one year from the time of the burn injury at 2-3 months post burn when deemed appropriate for pressure therapy, and have been evaluated as an appropriate candidate by a surgeon involved in this study for inclusion.
* subjects can be included up to one year post burn if referred from another treatment facility.
* no skin conditions that could potentially have an adverse effect on wound healing
* all race/ethnic groups
* children/guardians or significant others ability to speak English or Spanish and respond to study questionnaires.

Exclusion Criteria:

* subjects less than 9 years old as this age group is more fragile.
* subjects with no second degree burn to thigh and or trunk
* subjects with chemical burns
* subjects at low risk for hypertrophic scaring (wounds that demonstrate fading erythema at 9-12 weeks and wounds that are healed at less than 3 weeks are at low risk for hypertrophic scaring). Vancouver scar scale pigmentation rating of 0 or 1, vascularity rating of 0 or 1.
* TBSA greater than 50% as massive burns will confound results.
* potential life threatening injuries which would confound the effects of laser treatment and complicate sequential administration of therapy (e.g. shock,sepsis,inhalation therapies, brain injury).
* subjects with other inclusion criteria not met and evaluation by surgeon negative for inclusion in study.
* children/guardians or significant others inability to speak English or Spanish and respond to questionnaires.
* SUBJECTS WITH DOCUMENTED HYPERSENSITIVITY/ALLERGY TO AQUAPHOR,LIDOCAINE OR ANY OF THEIR COMPONENTS.

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-03 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Matching Assessment of Scars and Photographs | 12 months after the first laser procedure is completed
  This scar assessment tool uses a set of reference photographs, a numeric scale, and location technique to measure change over time of a burn scar. This tool will assist us in determining the comparative merits of laser treatments. It is portable and inexpensive.

SECONDARY OUTCOMES:
Burn Outcomes Questionnaire | Baseline completion after enrollment and again at 1st,2nd, 3rd, 4th,5th and 6th outpatient visits.
  The ABA/SHC Burn Outcomes Questionnaires are burn and age specific. Questions include those about itch, appearance and function; all elements of daily life that may be compromised by hypertrophic scars.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Donelan, MD, Principal Investigator — Shriners Hospitals for Children-Boston MA USA
Locations (1):
- Shriners Hospitals for Children, Cincinnati, Ohio, United States